CLINICAL TRIAL: NCT02102386
Title: Monitoring Brain Perfusion and Cerebral Oximetry in Carotid Endarterectomy Surgeries
Acronym: CerOx
Status: Terminated | Type: Observational
Why Stopped: Technical issues with the device under study. Sponsor terminated.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, kangrga, Clinical Chief Director, Abdominal Organ Transplant, Washington University School of Medicine
Other Study IDs: 201312041
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Carotid Endarterectomy
Keywords: elective; carotid endarterectomy surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CerOx: Patients will be monitored using the CerOx monitor. Probes will be attached bi-laterally in the OR to the forehead.

SUMMARY:
The goal of this study is to demonstrate Or-Nim's CerOx monitor ability to monitor changes in cerebral blood flow and oximetry during CEA surgery.

Procedures include:

Screening:

ECG, blood draw, neurological assessment, NIHSS

study: CerOX and TCD clock during CEA procedure, data collection from the medical record/monitors, neurological assessment, NIHSS

30 day follow-up

ELIGIBILITY:
Patients scheduled to undergo a CEA procedure that have consented to participate in the study will be included in this observational study.

Research Subjects: Indications for monitoring include patients scheduled for CEA that comply with the inclusion and exclusion criteria.

Inclusion Criteria

To be considered eligible to participate in this study, a patient must meet the inclusion criteria listed below:

1. Consenting patients over 18 years, undergoing elective carotid endarterectomy at Barnes Jewish Hospital.

Exclusion Criteria

To be eligible for entry into the study, the patient must not meet any of the exclusion criteria listed below:

1. Emergency surgery
2. National Institute of health Stroke Scale (NIHSS) score >=10
3. Sub-cutaneous hematoma at the ipsilateral intended area of the CerOx probe location.
4. Laceration or scalp injury at the ipsilateral intended area of the CerOx probe location which contraindicates placement of the adhesive on the skin.
5. Patient with implants located in the intended area of the CerOx probe location.
6. Prisoners
7. Non-consenting patient Or non-participating surgeon schedule of assessments and procedures
8. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective carotid endarterectomy at Barnes Jewish Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
compare cerebral perfusion and Oximetry changes to arterial blood pressure and trans-cranial doppler velocity changes | up to 3 hours
  compare cerebral perfusion and Oximetry changes to arterial blood pressure and trans-cranial doppler velocity changes

SECONDARY OUTCOMES:
to compare cerebral perfusion and oximetry changes to non-invasive cardiac output, and systemic vascular resistances changes. | up to 3 hours
  to compare cerebral perfusion and oximetry changes to non-invasive cardiac output, and systemic vascular resistances changes.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Kangrga, MD, PhD, Principal Investigator — Washington Univesity School of Medicine; Andrea Vannucci, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States